CLINICAL TRIAL: NCT01634815
Title: Evaluation of Local Capillary Blood Lactate in Chronic Critical Ischemia of Lower Limb Before and After Revascularization.
Acronym: ELIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5244
Record Dates: First submitted 2012-07-02; First posted 2012-07-06 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Chronic Critical Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lactate group (Experimental)
  Interventions: Procedure: The Edge

INTERVENTIONS:
Procedure: The Edge — measuring blood lactate

SUMMARY:
Evaluation of a new biological criterion, the local capillary blood lactates to optimize the management of patients with chronic critical ischemia requiring revascularization fast. Potential use in terms of capillary blood lactate as a diagnostic indicator of recurrent ischemia in a limb revascularized.

ELIGIBILITY:
Inclusion Criteria:

* Ischemia Chronic critical lower limb revascularization procedure requiring fast.
* Written consent informed patient age greater than or equal to 18

Exclusion Criteria:

* Presence of an inflammatory or infectious (erysipelas) in the ischemic member.
* Patients at risk for diabetic foot ie, as defined by the HAS (preventing diabetic foot, 2007)

  * presence of sensory neuropathy, and / or
  * foot deformities (hallux valgus, hammer toes or claw, prominence of the metatarsal heads), and / or
  * history of foot ulceration, and / or
  * antecedent of one of these factors (ie antécedant diabetic foot).
* Necrosis of the toes.
* Participation in another clinical research protocol.
* Presence of peripheral arterial disease in the bilateral upper limbs.
* Patient in shock whatever the cause.
* Presence of hepatic failure.
* Too impaired general condition (bedridden, dementia, ...)
* Refusal of the patient to participate in the study
* Protected patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02-04 (Actual); Primary Completion 2015-08-21 (Actual); Study Completion 2015-08-21 (Actual)

PRIMARY OUTCOMES:
Report Capillary blood lactate To Finger Capillary blood lactate (LCO / LCD) | 48 hours
  Report Capillary blood lactate To Finger Capillary blood lactate (LCO / LCD) before revascularization of the lower limb in chronic critical limb ischemia (considered positive if> 2).

SECONDARY OUTCOMES:
The decrease in the ratio LCO/LCD | 48 hours
  The decrease in the ratio LCO / LCD in the immediate aftermath of revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Diemunsch, MD, Principal Investigator — not affiliated
Locations (2):
- France (2):
  - Clinique de l'Orangerie, Strasbourg
  - Hôpitaux Universitaires de Strasbourg, Service d' Anesthésie Réanimation Chirurgicale, Strasbourg